CLINICAL TRIAL: NCT04310293
Title: Novel Therapy for Poor Responders Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, medical director, Al Baraka Fertility Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kamal-Rageh
Record Dates: First submitted 2020-03-08; First posted 2020-03-17 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Poor Ovarian Response
Keywords: IVF; POOR RESPONDERS; GROWTH HORMONE
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POOR RESPONDERS (Other): poor responders low AMH LOW AFC
  Interventions: Other: Femara,Grotwth hormone,HMG

INTERVENTIONS:
Other: Femara,Grotwth hormone,HMG — NOVEL THERAPY

SUMMARY:
Unfortunately for some infertile women, gonadotrophin administration results in a desultory ovarian response. While this is commonly due to diminished ovarian reserve, as indicated by advanced age and/or elevated basal day 3 FSH concentrations, a subset of these patients are <41 years old and have normal FSH concentrations.

To overcome this problem several strategies have been reported, with limited success.

With approval of the Board, 100 women with a history of previous poor response to vigorous gonadotrophin stimulation. All with AFC ≤3, AMH;≤0.5 and they give only ≤3 oocytes in their previous cycles will be included in this study using this new protocol: clomiphene citrate 150 for 7 days starting on DAY2, associated with HMG 300 IU & Groth hormone 8 units in alternating days (i.e.; HMG on D2,4,6,8 while GH on D3,5,7,9) then folliculomonitoring will be started on D9, then Antagonist may be added till triggering then will see the response compared to their own ovarian response before

DETAILED DESCRIPTION:
Unfortunately for some infertile women, gonadotrophin administration results in a desultory ovarian response. While this is commonly due to diminished ovarian reserve, as indicated by advanced age and/or elevated basal day 3 FSH concentrations, a subset of these patients are <41 years old and have normal FSH concentrations.

To overcome this problem several strategies have been reported, with limited success.

With approval of our Board, 100 women with a history of previous poor response to vigorous gonadotrophin stimulation. All with AFC ≤3, AMH;≤0.5 and they give only ≤3 oocytes in their previous cycles will be included in this study using this new protocol: clomiphene citrate 150 for 7 days starting on DAY2, associated with HMG 300 IU & Groth hormone 8 units in alternating days (i.e.; HMG on D2,4,6,8 while GH on D3,5,7,9) then folliculomonitoring will be started on D9, then Antagonist may be added till triggering then will see the response compared to their own ovarian response before in their previous trials

ELIGIBILITY:
Inclusion Criteria:

* All with AFC ≤3,
* AMH;≤0.5
* and they give only ≤3 oocytes in their previous cycles

Exclusion Criteria:

-

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
NUMBER OF OOCYTES | 2 weeks
  NUMBER

CONTACTS AND LOCATIONS:
Locations (1):
- Al-BARAKA FERTILITY HOSPITAL, Manama, Bahrain

IPD SHARING:
Plan to Share IPD: Undecided